CLINICAL TRIAL: NCT07279571
Title: GYN-AIDE: Gynecologic Oncology Navigation Through AI-Driven Education
Status: Not yet recruiting | Type: Observational
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 5U-25-1; NCI-2025-03594 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); UP-25-00331; 5U-25-1 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2025-11-20; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Patients complete a survey on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study
  Other Names: Non-Interventional Observational Study; Noninterventional (Observational) Study

SUMMARY:
This study seeks to understand how endometrial cancer patients get medical information about cancer care and their satisfaction with those health-seeking methods. It also assesses patient interest in using an artificial intelligence educational resource.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine how patients with endometrial cancer in the LA General Medical Center gynecologic oncology clinic currently obtain information about endometrial cancer care, and patient satisfaction with those health-seeking methods.

OUTLINE: This is an observational study.

Patients complete a survey on study.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the LA General gynecologic oncology clinic
* Age 18 years or older
* Biopsy-proven diagnosis of endometrial cancer
* Willing and able to provide informed consent

Exclusion Criteria:

* Patients who do not speak English or Spanish
* Patients who do not provide informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the LA General gynecologic oncology clinic with a biopsy-proven diagnosis of endometrial cancer.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-06-09 (Estimated); Study Completion 2026-06-09 (Estimated)

PRIMARY OUTCOMES:
Current medical resources used by patients and perceived relative importance of those resources | Up to 1 year
  Will be analyzed using a qualitative description with a potential subgroup analysis of current medical resources based on various demographic information.

SECONDARY OUTCOMES:
Demographics of patients | Up to 1 year
  Will be analyzed using a qualitative description of the demographics of patients involved in this specific study.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyue M Guo, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California